CLINICAL TRIAL: NCT04727853
Title: A Multicenter, Open-label, Single-arm Phase 2 Study of Irinotecan Liposome Injection in Patients With Small Cell Lung Cancer (SCLC) Who Have Progressed After Platinum-based First-line Therapy
Brief Title: Study of Irinotecan Liposome Injection as Second-line Regimen in Patients With Small Cell Lung Cancer (SCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE072-CSP-001
Record Dates: First submitted 2021-01-18; First posted 2021-01-27 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Small Cell Lung Cancer (SCLC)
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — irinotecan sucrosofate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- irinotecan liposome injection (Experimental): Patients will receive irinotecan liposome injection at 70 mg/m^2 intravenously, over 90 min on Days 1 of every 14-day cycle.
  Interventions: Drug: irinotecan liposome injection

INTERVENTIONS:
Drug: irinotecan liposome injection — Drug: irinotecan liposome injection

SUMMARY:
This study is a multicenter, open-label, single-arm phase 2 study of irinotecan liposome injection in patients with small cell lung cancer (SCLC) who have progressed after platinum-based first-line therapy. Subjects will receive irinotecan liposome injection until progression or unacceptable toxicity.

DETAILED DESCRIPTION:
Patients with small cell lung cancer who have progressed after platinum-based first-line therapy will be enrolled in this study. Patients will receive irinotecan liposome injection at 70 mg/m^2 intravenously, over 90 min on Days 1 of every 14-day cycle until progression or unacceptable toxicity. Imaging assessments will be conducted every three cycles to evaluate the preliminary efficacy of irinotecan liposome injection as second-line regimen in patients with SCLC.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age. Males or females.
2. Histopathologically or cytologically confirmed small cell lung cancer.
3. At least one measurable lesion as defined by RECIST V1.1 guidelines. A previously irradiated lesion may be counted as a measurable lesion only if there is a clear sign of progression since the irradiation.
4. Must have recurrence or progression after platinum-based, first-line chemotherapy or chemoradiation therapy for the treatment of SCLC.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy >3 months.
7. Recovered from the effects of any prior chemotherapy, surgery, radiotherapy or other anti-neoplastic therapy (recovered to no more than Grade 1 of CTCAE 5.0 criteria or baseline, with the exception of alopecia or other toxicity without safety concerns by the investigators' judgment).
8. Patient should not receive blood transfusion or supportive care (eg. EPO, G-CSF or others) within 14 days before the initiate dose, and laboratory test should meet the following criteria: neutrophile count (ANC) ≥1.5×10^9/L, platelet count ≥100×10^9/L, hemoglobin ≥90 g/L or ≥5.6 mmol/L, serum creatinine ≤1.5×ULN and creatinine clearance rate ≥30 mL/min, total bilirubin ≤1×ULN, AST and ALT ≤2.5×ULN (for patients with liver metastasis: ≤5×ULN)
9. Female or male patient of childbearing age must agree to take effective contraception for the duration of treatment plus six months post-treatment completion; female patient must have a negative serum pregnancy test within 7 days before enrollment and must not be lactating female.
10. Able to understand and provide an informed consent.

Exclusion Criteria:

1. Patients with large cell neuroendocrine lung carcinoma or combined small cell lung carcinoma.
2. Patients with history of immunotherapy-induced colitis or pneumonia, confirmed by clinical assessment and/or biopsy.
3. Patients with central Nervous System (CNS) metastasis meet any of the following criteria: a) Patient who have developed new or progressive brain metastasis following cranial radiation; b) Patients with the symptomatic Central Nervous System (CNS) metastasis who have used cortisol, radiotherapy, dehydration drugs, etc. to control symptoms in the past two weeks; c) Patients with carcinomatous meningitis; d) Patients with brain stem (midbrain, pons, medulla oblongata) or spinal cord metastasis.
4. Uncontrolled third lacunar effusion, not suitable for enrollment by investigator's assessment.
5. Previous malignancies in the past five years (except for basal cell carcinoma, squamous cell carcinoma, superficial bladder carcinoma, local prostate carcinoma, carcinoma in situ of cervical, or of others that have been radically resected and have not recurred).
6. Patients who have received any of the following treatments, a) Patients who have received prior topoisomerase I inhibitor treatment, including irinotecan or other investigational agents; b) Patients who have used any antibody-drug conjugates or molecular targeted preparation alone or in combination setting; c) Patients who have received more than one line of immunotherapy (immunotherapy in first-line as single or combination is permitted).
7. Concomitant use of strong CYP3A4 inducers within 2 weeks or strong CYP3A4 inhibitors or strong UGT1A1 inhibitors within 1 week of the first dose of the study drug.
8. Patients who have received any chemotherapy, biological therapy, endocrinotherapy, immunotherapy or investigational therapy within 4 weeks (5 half-lives of the agent, whichever is longer) of the first dose of the study drug, or local palliative radiotherapy or Chinese herbal medicine with anti-tumor indications within 2 weeks of the first dose of the study drug.
9. Any major surgery or severe trauma within 4 weeks of the first dose, not including biopsy.
10. Severe cardiovascular disease within 6 months prior to enrollment.
11. Severe pulmonary disease within 6 months prior to enrolment, such as interstitial pneumonia, pulmonary fibrosis, radiation induced pneumonitis requiring steroid therapy, and other moderate and severe lung diseases which affect lung function.
12. Uncontrolled active bleeding or known hemorrhagic constitution.
13. Any active infection, in the investigator's opinion, would increase the risk or have an influence on the result of the study, such as acute bacterial infection, tuberculosis, active hepatitis B/C, or HIV infection.
14. Known hypersensitivity to any of the components of irinotecan liposome injection, or other liposomal products.
15. Clinically significant gastrointestinal disorder, including hepatic disorders, bleeding, inflammation, occlusion, or diarrhea > grade 1.
16. History of explicit neurological or psychiatric disorders, including epilepsy or dementia.
17. Pregnant or lactating female.
18. Patient is not suitable for the study in the investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From date of first dose until the date of first documented progression, assessed up to 24 months
  ORR was defined as the proportion of patients who achieved partial response or complete response according to RECIST V1.1 guidelines.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  from date of the first dose to date of the first documented disease progression (PD) per RECIST v1.1 or death due to any cause, whichever occurs first.
Overall survival (OS) | From date of first dose until the date of death from any cause , assessed up to 24 months
  from date of the first dose to date of death from any cause
Proportion of Patients with Symptom Improvement | date of the first dose to 30 days after permanent treatment termination
  Patient-reported EORTC-QLQ symptom scales
Incidence of treatment-emergent adverse events (AEs), serious adverse events (SAEs) and laboratory abnormalities | date of the first dose to 30 days after permanent treatment termination
  Incidence of AE, SAE and laboratory abnormalities

OTHER OUTCOMES:
PK parameters-Cmax | Cycle 1（each cycle is 14 days）
  Cmax of total, encapsuled and free irinotecan
PK parameters-AUC | Cycle 1（each cycle is 14 days）
  AUClast, AUCinf of total, encapsuled and free irinotecan
PK parameters-others | Cycle 1（each cycle is 14 days）
  tmax, tlast, t1/2 of total, encapsuled and free irinotecan

CONTACTS AND LOCATIONS:
Overall Officials: Yin Cheng, Professor, Principal Investigator — Jilin Provincial Tumor Hospital
Locations (1):
- Jilin Cancer Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No